CLINICAL TRIAL: NCT03458780
Title: Single Cell Transcriptomics for Characterizing the Human Immune Response to Yellow Fever Vaccination
Brief Title: Yellow Fever Immune Response at Single Cell Resolution
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Brad Rosenberg, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: BRO-0905; 5U19AI111825 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: yellow fever vaccine; immune response; droplet microfluidics single cell ("inDrop") RNA-Seq
MeSH Terms: interventions — Yellow Fever Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research Bloods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Yellow Fever Vaccine Participant: Healthy participants who receive the Yellow fever vaccine for travel and/or occupational risk will have peripheral blood samples collected longitudinally at time points selected for different immune events post-vaccination according to published studies (Day 0 baseline; Days: 3, 7, 14, and 42).
  Interventions: Drug: Yellow Fever Vaccine

INTERVENTIONS:
Drug: Yellow Fever Vaccine — Yellow Fever Vaccine .5 ml
  Other Names: YF-Vax

SUMMARY:
The immune system is composed of diverse cell types with different functions that act together in order to defend against infection. This pilot study will test a new technology for studying these many different cell types at very large numbers at the level of individual cells. This method will then be used to identify the cell types and functions important for the immune response to the highly protective yellow fever vaccine, which will improve our understanding of effective vaccine features.

DETAILED DESCRIPTION:
Vaccines have had monumental impact in reducing the mortality and morbidity of infectious disease. However, the underlying immune mechanisms that contribute to their effectiveness are incompletely understood. Transcriptomics (methods that measure the activity of thousands of genes) studies have identified key features of responses to vaccination(see references) and infection(see references). However, these experiments are typically performed on heterogeneous cell mixtures such as peripheral blood mononuclear cells (PBMC which include certain types of white blood cells) and therefore provide an aggregate measure of gene expression from the many different immune cells and their respective activities in the mixture. Such results can obscure important biological information, particularly in minor subsets of active cells. Establishing a method for immune transcriptomics at single cell resolution would be a highly significant advance and enable more informative and functionally relevant systems immunology studies with commonly used sample types (i.e. PBMC). Applying this high-resolution approach to Yellow Fever Vaccine (YFV), an exceptionally effective vaccine, is likely to identify unappreciated mechanisms that contribute to protective immunity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 59 years old
* Volunteers who have not received a vaccination within 30 days of the YFV and do not anticipate to receive a vaccination within 30 days
* Volunteers who are seeking the YFV for either travel reasons or occupational risk
* Volunteers willing to undergo one screening visit, one visit to receive the YFV, and four post-vaccination visits
* Volunteers without medical conditions who are willing to give blood once for the development of the inDrop technique

Exclusion Criteria:

* Male or females under 18 or over 59 years of age
* Volunteers who received other vaccination less than 30 days prior to receiving the YFV
* Volunteers with acute or febrile disease
* Volunteers unable to return for the post vaccination follow-up visits
* Volunteers with an allergy to eggs, chicken proteins, gelatin, or other components of the Yellow Fever vaccine
* Participation in another clinical study of an investigational product currently or within the past 90 days, or expected participation during this study
* Is pregnant or lactating
* Volunteers with a history of yellow fever vaccination and/or infection
* Volunteers with a history of viral hepatitis and/or non-viral liver disease
* In the opinion of the investigators, the volunteer is unlikely to comply with the study protocol
* Immunosuppressed individuals as a result of cancer, transplantation, and or primary immunodeficiency
* Immunosuppressed individuals as a result of medications (such as high-dose systemic corticosteroids, alkylating drugs, antimetabolites, TNF-α inhibitors (e.g., etanercept), IL-1 blocking agents (e.g., anakinra), and other monoclonal antibodies targeting immune cells (e.g.,rituximab, alemtuzumab) and/or radiation
* Volunteers with thymus disorders (including myasthenia gravis, Di George syndrome, or thymoma) and/or history of thymectomy
* Individuals infected with HIV

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2016-08-22 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Feasibility and accuracy of inDrop RNA-Seq | up to 42 days post baseline visit
  The feasibility and accuracy of inDrop RNA-Seq for distinguishing different cell types will be assessed by comparing (for concordance) cell subset population frequency and distribution values determined by inDrop RNA-seq to cell subset population frequency and distribution values determined by flow cytometry immunophenotyping, the present "gold standard" technique.

SECONDARY OUTCOMES:
Utility of inDrop RNA-Seq | Days 0, 3, 7, 14, 42
  The utility of inDrop RNA-Seq for characterizing an immune response will be determined by measuring cell subset frequencies and gene expression profiles at single cell resolution over time following YFV.

CONTACTS AND LOCATIONS:
Overall Officials: Brad R Rosenberg, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Rockefeller University, New York, New York, United States

REFERENCES:
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Obermoser G, Presnell S, Domico K, Xu H, Wang Y, Anguiano E, Thompson-Snipes L, Ranganathan R, Zeitner B, Bjork A, Anderson D, Speake C, Ruchaud E, Skinner J, Alsina L, Sharma M, Dutartre H, Cepika A, Israelsson E, Nguyen P, Nguyen QA, Harrod AC, Zurawski SM, Pascual V, Ueno H, Nepom GT, Quinn C, Blankenship D, Palucka K, Banchereau J, Chaussabel D. Systems scale interactive exploration reveals quantitative and qualitative differences in response to influenza and pneumococcal vaccines. Immunity. 2013 Apr 18;38(4):831-44. doi: 10.1016/j.immuni.2012.12.008. PMID 23601689
- [Background] Tsang JS, Schwartzberg PL, Kotliarov Y, Biancotto A, Xie Z, Germain RN, Wang E, Olnes MJ, Narayanan M, Golding H, Moir S, Dickler HB, Perl S, Cheung F; Baylor HIPC Center; CHI Consortium. Global analyses of human immune variation reveal baseline predictors of postvaccination responses. Cell. 2014 Apr 10;157(2):499-513. doi: 10.1016/j.cell.2014.03.031. PMID 24725414
- [Background] Li S, Rouphael N, Duraisingham S, Romero-Steiner S, Presnell S, Davis C, Schmidt DS, Johnson SE, Milton A, Rajam G, Kasturi S, Carlone GM, Quinn C, Chaussabel D, Palucka AK, Mulligan MJ, Ahmed R, Stephens DS, Nakaya HI, Pulendran B. Molecular signatures of antibody responses derived from a systems biology study of five human vaccines. Nat Immunol. 2014 Feb;15(2):195-204. doi: 10.1038/ni.2789. Epub 2013 Dec 15. PMID 24336226
- [Background] Gaucher D, Therrien R, Kettaf N, Angermann BR, Boucher G, Filali-Mouhim A, Moser JM, Mehta RS, Drake DR 3rd, Castro E, Akondy R, Rinfret A, Yassine-Diab B, Said EA, Chouikh Y, Cameron MJ, Clum R, Kelvin D, Somogyi R, Greller LD, Balderas RS, Wilkinson P, Pantaleo G, Tartaglia J, Haddad EK, Sekaly RP. Yellow fever vaccine induces integrated multilineage and polyfunctional immune responses. J Exp Med. 2008 Dec 22;205(13):3119-31. doi: 10.1084/jem.20082292. Epub 2008 Dec 1. PMID 19047440
- [Background] Fourati S, Cristescu R, Loboda A, Talla A, Filali A, Railkar R, Schaeffer AK, Favre D, Gagnon D, Peretz Y, Wang IM, Beals CR, Casimiro DR, Carayannopoulos LN, Sekaly RP. Pre-vaccination inflammation and B-cell signalling predict age-related hyporesponse to hepatitis B vaccination. Nat Commun. 2016 Jan 8;7:10369. doi: 10.1038/ncomms10369. PMID 26742691
- [Background] Kwissa M, Nakaya HI, Onlamoon N, Wrammert J, Villinger F, Perng GC, Yoksan S, Pattanapanyasat K, Chokephaibulkit K, Ahmed R, Pulendran B. Dengue virus infection induces expansion of a CD14(+)CD16(+) monocyte population that stimulates plasmablast differentiation. Cell Host Microbe. 2014 Jul 9;16(1):115-27. doi: 10.1016/j.chom.2014.06.001. Epub 2014 Jun 26. PMID 24981333
- [Background] Suthar MS, Pulendran B. Systems analysis of West Nile virus infection. Curr Opin Virol. 2014 Jun;6:70-5. doi: 10.1016/j.coviro.2014.04.010. Epub 2014 May 20. PMID 24851811